CLINICAL TRIAL: NCT04026867
Title: Determining Effective Testing in Emergency Departments and Care Coordination on Treatment Outcomes (DETECT) for HCV
Brief Title: The DETECT HCV Linkage to Care Trial
Acronym: DETECT HCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jason Haukoos, Professor & Director of Research, Department of Emergency Medicine, Denver Health, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-2327; R01DA042982 (NIH)
Record Dates: First submitted 2019-06-27; First posted 2019-07-19 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-02

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinician Referral Only (Active Comparator): The Clinician Referral arm will serve as an "active control" and baseline standard of care. All individuals who test positive for HCV antibodies or are identified with untreated, active HCV will be informed of their result and receive the following information from their clinical care teams in the ED: (a) explanation of process and rationale for follow-up RNA testing; (b) delivery of simple posttest counseling (e.g., risk for liver disease, risks of transmission); and (c) provision of a list of insurance enrollment resources, as needed, along with (d) a list of HCV treatment providers and their contact information as provided in aftercare instructions. For new HCV diagnoses, patients will be instructed to access their electronic patient portal (MyChart) for their RNA test results or to call a designated results line. Post-testing counseling messages and follow-up instructions will be included on the patient discharge papers.
  Interventions: Other: Clinician Referral
- Clinician Referral + Linkage Navigation (Experimental): The Linkage Navigation arm will consist of an additional service layered onto clinician referral and will incorporate protocols from Antiretroviral Treatment and Access Studies (ARTAS). Individuals randomized to this intervention will be contacted by a linkage navigator either during the ED visit (if during business hours) or the following business day (if during non-business hours). If the navigator does not contact the patient at the time of ED visit, they will offer to meet with the patient in person or over the phone. For all individuals in this arm, a structured linkage navigation process will include motivational interviewing and (a) reiteration of posttest counseling messages, (b) assessment of the patient's needs for medical insurance and substance abuse treatment, c) assistance scheduling and/or rescheduling appointments for HCV treatment, and d) follow-up phone call after the first HCV treatment appointment and thereafter as needed up to 6 months after ED visit.
  Interventions: Other: Linkage Navigation; Other: Clinician Referral

INTERVENTIONS:
Other: Linkage Navigation — The Linkage Navigation arm will consist of an additional service layered onto clinician referral and will incorporate protocols from Antiretroviral Treatment and Access Studies (ARTAS), the most influential studies of HIV linkage-to-care to date.
  Arms: Clinician Referral + Linkage Navigation
Other: Clinician Referral — The Clinician Referral arm will serve as an "active control" and baseline standard of care.

SUMMARY:
This aim of the DETECT HCV linkage trial compares two linkage to care intervention strategies among (1) newly diagnosed HCV positive patients from the emergency department (ED) and (2) those patients who present to the ED with untreated active HCV. Patients who are positive for HCV and agree to be part of the study will be randomized to either clinician referral alone or clinician referral plus a linkage navigator.

DETAILED DESCRIPTION:
The investigators will perform a prospective pragmatic randomized effectiveness trial to compare 2 linkage-to-care strategies. Permuted block randomization with 2 strata (i.e., <40 years of age or active IDU [defined as IDU within 30 days], or ≥40 years of age without active IDU) and varying block sizes will be used to minimize imbalance, ensure appropriate numbers of patients in subgroups, and allow for efficient analyses. Allocation will be concealed by blinding block sizes and using the REDCap Randomization Module, a web-based platform to assign patients to arms (REDCap, Vanderbilt University, TN). Although patients will not be blinded to the interventions, they will be blinded to the outcomes. Also, a trained research assistant will perform all enrollment, including stratification and randomization. Clinical staff will not be blinded, however, to assignment.

ELIGIBILITY:
Inclusion Criteria:

* ED patients who test positive for HCV antibodies
* ED patients who have discharged and confirmatory RNA result is positive
* Clinically stable per screening nurse or physician assessment
* Able to provide consent
* ED patients with untreated active HCV confirmed by the electronic medical record

Exclusion Criteria:

* Younger than 18 years of age
* Prisoners
* Pregnant women
* Individuals that live out of state
* Unable to consent for care (e.g., altered mentation, critical illness or injury)
* Non English or Spanish speaking
* Have already participated in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Number of individuals who fill a prescription for Direct-Acting Antivirals (DAAs) for hepatitis C within 6 months of positive HCV RNA test (for new HCV diagnosis) or presenting at ED visit (for those identified with untreated, active HCV). | Within 6 months from time of HCV diagnosis (for new HCV diagnoses) or ED visit (for those identified with untreated, active HCV).
  The primary outcome will be the number of individuals with positive HCV RNA test who initiate HCV treatment within 6 months from the time of ED diagnosis (for new HCV diagnoses) or from time of ED visit (for those identified with untreated, active HCV). This will be verified by electronic medical record review.

SECONDARY OUTCOMES:
Number of individuals who attend an appointment with an HCV treatment provider within 6 months of positive HCV RNA test (for new HCV diagnoses) or ED visit (for existing HCV diagnoses). | Within 6 months from time of HCV diagnosis (for new HCV diagnoses) or ED visit (for existing HCV diagnoses)
  Measured by indication of a completed visit with an HCV treatment provider among those identified with active HCV. This will be verified by electronic medical record review.

OTHER OUTCOMES:
For individuals who self-identify as a person who injects drugs (PWID), the number of individuals who initiate substance use disorder services within 6 months of positive HCV RNA test (for new HCV diagnoses) or ED visit (for existing HCV diagnoses). | Within 6 months from time of HCV diagnosis (for new HCV diagnoses) or ED visit (for existing HCV diagnoses).
  Measured by indication of a completed visit with a substance use treatment provider. This will be verified via electronic medical record review.
Number of individuals who complete their full course of HCV treatment with DAAs within 6 months of positive HCV RNA test (for new HCV diagnoses) or ED visit (for existing HCV diagnoses). | Within 6 months from time of HCV diagnosis (for new HCV diagnoses) or ED visit (for existing HCV diagnoses).
  Measured by indication of completion of treatment with DAAs among those individuals identified with active HCV. This will be verified by electronic medical record review.
Number of individuals who have documented sustained virologic response 12 weeks after completing treatment with DAAs within 6 months of positive HCV RNA test (for new HCV diagnoses) or ED visit (for existing HCV diagnoses). | Within 6 months from time of HCV diagnosis (for new HCV diagnoses) or ED visit (for existing HCV diagnoses).
  Rates of sustained virologic response within 12 weeks (SVR12) will be measured by report of undetectable HCV RNA Nucleic Acid Amplification Test (NAAT) 12 weeks after completion of DAAs among those identified with active HCV. This will be verified by electronic medical record review.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rowan, MD, Principal Investigator — Denver Health; Jason Haukoos, MD, MSc, Principal Investigator — Denver Health
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rowan SE, Haukoos J, Kamis KF, Hopkins E, Gravitz S, Lyle C, Al-Tayyib AA, Gardner EM, Galbraith JW, Hsieh YH, Lyons MS, Rothman RE, White DAE, Morgan JR, Linas BP, Sabel AL, Wyles DL; DETECT Hep C Trials Investigators. The Determining Effective Testing in Emergency Departments and Care Coordination on Treatment Outcomes (DETECT) for Hepatitis C (Hep C) Linkage-to-Care Trial: rationale and design of an emergency department-based randomized clinical trial of linkage-to-care strategies for hepatitis C. Trials. 2023 Jan 27;24(1):63. doi: 10.1186/s13063-022-07018-w. PMID 36707909